CLINICAL TRIAL: NCT04312321
Title: Audiovisual Consultations by Paramedics With an Emergency Medical Service Physician in Low Urgency Events: Randomised Controlled Trial
Brief Title: Audiovisual Consultations in Prehospital Emergency Care: Randomised Controlled Trial
Acronym: Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O. (Other)
Responsible Party: Principal Investigator, Roman Sýkora, MD, Ph.D., Principal Investigator, Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Telemedicina_10/11/2019
Record Dates: First submitted 2020-01-29; First posted 2020-03-18 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Telemedicine; Emergency Medical Service
Keywords: Pre-hospital care; Audiovisual consultation; Non-transport; Low urgency

STUDY DESIGN:
Intervention Model Description: Low urgency emergency calls are randomised by call-taker of dispatching center to 3 groups: routine prehospital emergency care without optional phone call consultation (1), with mandatory phone call consultation with base physician (2), with mandatory audivisual consultation with base physician (3). Power analysis. Based on available data prior to the initiation of the study, 10% of patients after low acuity calls were treated on site. The hypothesis that the video consult would lead to doubling this percentage will be investigated. In order to have 80% probability to confirm this at p < 0.05, we would need 200 subjects per group. Planned interim analysis will be after 4 weeks of study (aprox. after 600 eligible cases) .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): CONTROL group: low urgency cases with routine operation of paramedic crew with optional consultation with a doctor over the phone.
- PHONE (Experimental): In the PHONE group, there will be a mandatory consultation of a doctor over the phone in all low urgency cases.
  Interventions: Device: Mandatory phone call consultation
- VIDEO (Experimental): In the VIDEO group, there will be a mandatory consultation of a doctor over the audiovisual consultation in low urgency cases
  Interventions: Device: Mandatory audiovisual consultation

INTERVENTIONS:
Device: Mandatory phone call consultation — Use of audio consultation (EMS crew smartphones, doctor smarphone) Smartphone (Xiaomi Redmi Note) and bluetooth handsfree headset (Jabra Talk)
  Other Names: mandatory phone consultation (via Czech mobile network provider O2 Czech, GSM); mandatory telephone consultation (via Czech mobile network provider O2 Czech, GSM)
  Arms: PHONE
Device: Mandatory audiovisual consultation — Smartphone (Xiaomi Redmi Note) and bluetooth handsfree headset (Jabra Talk) with installed Android application (VSee messenger, USA, HIPAA compliant software) for paramedic crews; personal computer (Windows 10) with desktop version of application VSee messenger for Windows and eqipped with webcamera (Logitech C922 PRO) and headset (Jabra Evolve 20) for consulting doctor.
  Other Names: Mandatory video conference consultation
  Arms: VIDEO

SUMMARY:
This study investigates safety and efficacy of the use of audiovisual consultations of emergency medical service (EMS) doctor by paramedics for low urgency events in areas covered with paramedic crews only from emergency medical service stations with distant access to hospital.

DETAILED DESCRIPTION:
The study will be realized on Karlovy Vary EMS areas covered with paramedic crews only from emergency medical service stations with distant access to hospital. Each call on emergency line during 6 weeks study period will be assessed for eligibility. If deemed as low urgency, the event will be randomised into 3 groups. CONTROL group: routine operation of paramedic crew with optional consultation with a doctor over the phone. In the PHONE group and in the VIDEO group, there will be a mandatory consultation of a doctor over the phone or by audiovisual constultation, respectively. The primary outcome of the study is the percent of patients treated on site without the need of hospital transfer. The secondary safety outcome is to evaluate repeated ambulance trips within 48 hours after the patient had been treated at home. Moreover, a qualitative analysis of subjective perception of the event by the patients, paramedic and consulting doctor using the Likert scales will be performed by survey at the end or immediately after the event.

ELIGIBILITY:
Each call on emergency line (in action radius of actual position of 11 of 19 Karlovy Vary EMS paramedic crews) will be assessed for eligibility by EMS call-taker in Karlovy Vary region.

Inclusion criteria are:

1. the call is evaluated as low urgency event (by criteria of Karlovy Vary EMS call-taker manual; the event is dedicated for paramedic crew only, without dispatchig doctor on site),
2. the case is determined for and will be served by one of 11 for study dedicated of total 19 paramedic crews in Karlovy Vary EMS,
3. dedicated doctor of Karlovy Vary EMS will be available for consultation during his shift.

Exclusion criteria are:

1. need for escalation of the care: paramedics' requirement for the doctor to arrive at the scene of intervention,
2. consulting doctor is not available for the study at the moment of randomisation,
3. consultation with other than trained and for study dedicated doctors,
4. patient - crew language barrier,
5. study refusal by the patient or legal representative, or refusal of audiovisual consultation,
6. technical, logistic or other (agressive patient, patient detained by police) problems evaluated by paramedic crew (not to conduct a study in PHONE and especially VIDEO group)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Non-transport of low urgency EMS case to hospital | until 200 cases per group are collected, estimated time 6-8 weeks from the beginning of the study
  Based on Karlovy Vary EMS audit data, there is 10% of low urgency cases treated and left on site by paramedics so far. So the primary outcome is to evaluate the rate of non-transports in common daily routine, when the doctor provides phone call consultation on request of paramedics (based on Karlovy Vary EMS protocol) to mandatory phone call consultation and audiovisual consultation with a EMS doctor. Therefore, the primary objective is to evaluate potential benefit audiovisual consultation with EMS doctor on the rate of patients left at home after treatment on site by paramedics.

SECONDARY OUTCOMES:
The rate of repeated trips within 48 hours after the patient had been treated at home. | until 200 cases per group are collected, estimated time 6-8 weeks from the beginning of the study
  The co-primary safety outcome was repeated EMS trip within 48 hours after the patient had been treated at home. This outcome can confirm and compare the safety among study groups.

OTHER OUTCOMES:
Qualitative analysis of subjective perception of phone call and audivisual consultation. | until 200 cases per group are collected, estimated time 6-8 weeks from the beginning of the study
  This analysis of subjective perception of each event in all 3 groups will be evaluated. The inevstigators will use Likert scales (1-excellent, 2-good, 3-sufficient, 4-insufficient) to compare phone and audivisual consultation in following parameters: clinical information transfer, situational context, safety of care. Surveys have to be filled and the patient opinion should be asked at the and of an transport or befere the crew leaves the patient on site. The EMS doctor will fill the survey immediately after the phone or audiovisual consultation is provided.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Smetana, MD, Study Director — Zdravotnická záchranná služba Karlovarskeho kraje, PO
Locations (1):
- Zdravotnická záchranná služba Karlovarského kraje, p.o., Karlovy Vary, Karlovarský kraj, Czechia